CLINICAL TRIAL: NCT00838318
Title: Colorectal Cancer (CRC) Screening in First-Degree Relatives (FDRs) of Hispanic CRC Patients
Brief Title: Colon Cancer Screening in First-Degree Relatives of Hispanic Colorectal Cancer (CRC) Patients
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2004-0039
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Colorectal Cancer
Keywords: Colorectal CancerScreening; CRC; Hispanic; CRC Patients; First-Degree Relatives; FDRs; Interviews; Colorectal cancer screening; CRCS; Key Informants
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Arm 1 Hispanic CRC Patients
  Interventions: Behavioral: Interview
- Arm 2 FDRs of Hispancic CRC Patients: First-Degree Relatives (FDRs) of Hispanic CRC Patients
  Interventions: Behavioral: Interview
- Arm 3 Key Informants: Key informants from Houston Hispanic Health Coalition.
  Interventions: Behavioral: Interview

INTERVENTIONS:
Behavioral: Interview — Audiotaped Phone Interview/Survey, 30 - 45 minutes.

SUMMARY:
Primary Objectives:

1. To evaluate knowledge, beliefs, attitudes and values that influence perceptions and utilization of colorectal cancer screening (CRCS) among first-degree relatives of Hispanic CRC patients.
2. To assess factors influencing Hispanic CRC patients' communication of CRC risk and screening information to their FDRs.

Secondary Objective:

1) To establish the feasibility of recruiting Hispanic CRC patients and their FDRs from the institutional patient database and/or MDACC clinics.

DETAILED DESCRIPTION:
CRC PATIENTS AND THEIR FDRS:

You will be asked to complete a questionnaire by telephone interview. The study researcher who calls you will ask for your permission to audiotape the interview. The questionnaire asks about your awareness of screening tests for colorectal cancer, your family's past use of these screening tests, your attitudes toward colorectal cancer screening, and how you discuss colorectal cancer risk and screening with your family and health care providers. Some demographic information also will be collected (such as your age or marital status). The questionnaire will take between 30 and 45 minutes to complete.

Your answers to the questions and your personal information will be kept strictly confidential. Your questionnaire answers will be identified with a code number, rather than a name, so that you cannot be identified. Audiotaped recordings will be destroyed after all the data have been collected and studied (no longer than 5 years).

This is an investigational study. Up to 60 colorectal cancer patients and their close relatives may be enrolled in the study. All will be enrolled at M. D. Anderson.

KEY INFORMANT:

You will be asked to complete a psychosocial interview either in person or by telephone. The study staff member interviewing you will ask you for permission to audiotape the interview. You will be asked to review the interview guides for colorectal cancer patients and their first degree relatives (FDRs), and provide feedback about them. The interviewer will ask for your opinions about Hispanics' awareness and understanding of colorectal cancer screening. You will also be asked for your opinion about cultural beliefs and practices that may influence participation in colorectal cancer screening. The interview will take between 30 and 45 minutes to complete.

Your answers to the questions and your personal information will be kept strictly confidential. Your questionnaire answers will be identified with a code number, rather than a name, so that you cannot be identified. Audiotaped recordings will be destroyed after all the data have been collected and studied (no longer than 5 years).

This is an investigational study. Up to 15 key informants may be enrolled in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Key Informants: Persons will be identified as potentially eligible key informants if they are: 1) members of the Houston Hispanic Health Coalition, or if they are identified through the Houston Hispanic Health Coalition as having professional expertise relevant to this study. 2) Able to speak English or Spanish. 3) Able to provide informed consent.
2. CRC Patients: Eligibility criteria include: 1) Living MDACC patients with a personal history of colorectal adenocarcinoma (diagnosed as local or regional disease), who are between the ages of 18 and 60 years, who are identified as Hispanic/Latino, and who have living first degree relatives (siblings or children) between the ages of 40 and 70. 2) Able to provide informed consent. Eligible persons may speak either English or Spanish.
3. First-degree relatives (FDRs): Eligibility criteria include: 1) First-degree relatives (siblings and children) of the MDACC CRC cancer patients who are recruited to this study, who are 40 to 70 years of age. 2) Able to provide informed consent. Eligible persons may speak either English or Spanish.
4. Note: As described in the above inclusion criteria, this protocol involves recruiting and interviewing of key informants, CRC patients, and eligible first-degree relatives (FDRs) of CRC patients for three phases of the study.

Exclusion Criteria:

1. CRC Patients: CRC patients will be excluded if they have a history of a known hereditary CRC syndrome (e.g., HNPCC, familial polyposis) or inflammatory bowel disease (e.g., ulcerative colitis or Crohn's disease), or were diagnosed with distant metastases.
2. First degree relatives: FDRs of eligible CRC patients will be excluded if they have a history of a known hereditary CRC syndrome (e.g., HNPCC, familial polyposis) or inflammatory bowel disease (e.g., ulcerative colitis or Crohn's disease), or have a personal history of cancer (except non-melanoma skin cancer) or polyps.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Key Informants from Houston Hispanic Health Coaltion having professional expertise relevant to this study; MDACC Hispanic/Latino CRC Patients, age 18 - 60 years with first degree relatives between age 40 - 70; First-degree relatives (siblings and children) of the MDACC CRC cancer patients recruited to this study, who are aged 40 - 70 years.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2004-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To look at the knowledge, beliefs, and attitudes toward screening for colorectal cancer among Hispanic colorectal cancer patients and their close relatives. | 5 Years

SECONDARY OUTCOMES:
To study how these families communicate with each other and health care providers about colorectal cancer risk and screening. | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Susan Peterson, PhD, MPH, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org